CLINICAL TRIAL: NCT00421863
Title: Italian Study on the Cardiovascular Effects of Systolic Blood Pressure Control - CARDIOSIS Study
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Heart Care Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: C 33
Record Dates: First submitted 2007-01-12; First posted 2007-01-15 (Estimated); Last update posted 2021-02-03 (Actual); Status verified 2013-03

CONDITIONS: Hypertension
Keywords: hypertension; systolic blood pressure
MeSH Terms: conditions — Hypertension | interventions — Ramipril; Telmisartan; Amlodipine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intensive Strategy (Other)
  Interventions: Drug: Triatec 10 mg; Drug: Triatec HCT 5; Drug: Lasix 25; Drug: Micardis 80 mg; Drug: Micardis plus 80/12.5; Drug: Catapresan TTS 2; Drug: Norvasc 10 mg; Drug: Triatec 5 mg; Drug: Pluscor
- Usual Strategy (Other)
  Interventions: Drug: Triatec 10 mg; Drug: Triatec HCT 5; Drug: Lasix 25; Drug: Micardis 80 mg; Drug: Micardis plus 80/12.5; Drug: Catapresan TTS 2; Drug: Norvasc 10 mg; Drug: Triatec 5 mg; Drug: Pluscor

INTERVENTIONS:
Drug: Triatec 10 mg — Use and dosage according to physician judgement, concomitant treatment assumed and randomization arm (Intensive Strategy vs. Usual Strategy).
Drug: Triatec HCT 5 — Use and dosage according to physician judgement, concomitant treatment assumed and randomization arm (Intensive Strategy vs. Usual Strategy).
Drug: Lasix 25 — Use and dosage according to physician judgement, concomitant treatment assumed and randomization arm (Intensive Strategy vs. Usual Strategy).
Drug: Micardis 80 mg — Use and dosage according to physician judgement, concomitant treatment assumed and randomization arm (Intensive Strategy vs. Usual Strategy).
Drug: Micardis plus 80/12.5 — Use and dosage according to physician judgement, concomitant treatment assumed and randomization arm (Intensive Strategy vs. Usual Strategy).
Drug: Catapresan TTS 2 — Use and dosage according to physician judgement, concomitant treatment assumed and randomization arm (Intensive Strategy vs. Usual Strategy).
Drug: Norvasc 10 mg — Use and dosage according to physician judgement, concomitant treatment assumed and randomization arm (Intensive Strategy vs. Usual Strategy).
Drug: Triatec 5 mg — Use and dosage according to physician judgement, concomitant treatment assumed and randomization arm (Intensive Strategy vs. Usual Strategy).
Drug: Pluscor — Use and dosage according to physician judgement, concomitant treatment assumed and randomization arm (Intensive Strategy vs. Usual Strategy).

SUMMARY:
Multicenter, prospective, randomised, open study comparing the effect of the following two strategies in hypertensive subjects > 55 years and poorly controlled (systolic blood pressure >= 150 mmHg) by antihypertensive treatment:

* usual strategy: reduction of systolic blood pressure to below 140 mmHg, independently of diastolic blood pressure levels;
* intensive strategy: reduction of systolic blood pressure to below 130 mmHg, independently of diastolic blood pressure levels.

During the initial run in period two qualifying visits at distance of 7-14 days will be carried out to establish whether blood pressure remains uncontrolled (systolic blood pressure >=150 mmHg)by current drug treatment. At the end of the second visit eligible patients will be admitted to the study and the following examinations will be carried out: clinical visit, routine laboratory tests, 12-lead ECG. At this point eligible patients will be randomised to one of the two blood pressure goals outlined above.

Subsequent clinical visits will be carried out at 4 month-intervals up to the end of the study (4, 8, 12, 16, 20, 24 months).

DETAILED DESCRIPTION:
Study partially sponsored by: Boehringer Ingelheim, Sanofi-Aventis, Pfizer

ELIGIBILITY:
Inclusion Criteria:

* written informed consent to the study
* age >= 55 years at randomization. There is no upper age limit
* systolic blood pressure >= 150 mmHg in 2 visits at distance of 7-14 days, irrespective of diastolic pressure. Duration of treatment before visit 1 must be at least 12 weeks
* at least one additional risk factor including the following:
* current cigarette smoking
* total cholesterol >= 20 mmg/dl, or High Density Lipoproteins (HDL) < 40 mg/dl, or Low Density Lipoproteins (LDL) cholesterol >= 130 mg/dl
* family history of cardiovascular disease in male first degree relative < 55 years or female first degree relative < 65 years
* previous TIA or stroke
* previous coronary artery disease
* history of peripheral occlusive arterial disease (claudication intermittens associated with angiographic or echographic evidence of > 60% stenosis)

Exclusion Criteria:

* diabetes (fasting glucose > 125 mg/dl in two samples or ongoing diabetic treatment)
* renal failure, defined by a serum creatinine > 2.0 mg/dl
* chronic atrial fibrillation or flutter
* clinically significant hepatic or hematological disorders, alcoholism, drug addiction
* causes precluding ECG interpretation for LVH: complete right or left bundle block, Wolff-Parkinson-White syndrome, previous Q-wave myocardial infarction
* any disease causing reduced life expectancy
* unwilling to participate
* significant (more than traces of) valvular heart disease

Min Age: 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1111 (Actual)
Dates: Start 2005-02; Primary Completion 2009-01 (Actual); Study Completion 2009-01 (Actual)

PRIMARY OUTCOMES:
changes in Left Ventricular Hypertrophy (LVH) at Electro Cardio Gramme (ECG). | 0, 12, 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Paolo Verdecchia, MD, Study Chair — Ospedale Silvestrini - Perugia
Locations (45):
- Italy (45):
  - Ospedale N. Melli, San Pietro Vernotico, Brindisi
  - Ospedale Civile Mellini, Chiari, BS
  - Ospedale Civile G. Chidichimo, Trebisacce, Cosenza
  - Istituto Neuromed, Pozzilli, Isernia
  - Presidio Ospedaliero F. Ferrari, Casarano, Lecce
  - Nuovo Ospedale Versilia, Lido di Camaiore, Lucca
  - Ospedale Civile, Castiglione del Lago, Perugia
  - Ospedale Civile Beato Giacomo Villa, Città della Pieve, Perugia
  - Presidio Ospedaliero Città di Castello, Città di Castello, Perugia
  - Ospedale Civile, Gubbio, Perugia
  - Presidio Ospedaliero, Todi, Perugia
  - Ospedale Silvestrini, Perugia, PG
  - Ospedale Civile, Sacile, Pordenone
  - Ospedale Scillesi D'America, Scilla, Reggio Calabria
  - Ospedale Civile, Thiesi, Sassari
  - Presidio Ospedaliero, Poggibonsi, Siena
  - Ospedale Civile S. Antonio Abate, Erice, Trapani
  - Ospedale S. Antonio, San Daniele del Friuli, Udine
  - Ospedale Generale Regionale, Aosta
  - Azienda Ospedaliera G. Rummo, Benevento
  - Spedali Civili, Brescia
  - Azienda Ospedaliera G. Brotzu - S. Michele, Cagliari
  - Ospedale S. Elia, Caltanissetta
  - Ospedale Garibaldi-Nesima, Catania
  - Azienda Ospedaliera Mater Domini, Catanzaro
  - Ospedale Clinicizzato Santissima Annunziata, Chieti
  - Istituti Ospitalieri, Cremona
  - Dimi - Disem, Genova
  - Ospedale Generale Provinciale, Gorizia
  - Policlinico Universitario Federico II, Napoli
  - Azienda Ospedaliera di Perugia, Perugia
  - Spedali Riuniti, Pistoia
  - Ospedale Civile, Ragusa
  - Ospedali Riuniti G. Melacrino F. Bianchi, Reggio Calabria
  - Ospedale San Filippo Neri, Roma
  - CTO, Roma
  - Ospedlae San Camillo, Roma
  - Ospedale San Camillo, Roma
  - Ospedale San Giovanni, Roma
  - Policlinico Universitario, Sassari
  - Azienda Ospedaliera, Syracuse
  - Azienda USL 4 Terni, Terni
  - Ospedale San Vito, Torino
  - Casa di Cura Villa Bianca, Trento
  - Ospedale Belcolle, Viterbo

REFERENCES:
- [Background] Cardio-Sis Study Group. Randomized study of traditional versus aggressive systolic blood pressure control (Cardio-Sis): rationale, design and characteristics of the study population. J Hum Hypertens. 2008 Apr;22(4):243-51. doi: 10.1038/sj.jhh.1002313. Epub 2007 Nov 29. PMID 18046432
- [Result] Verdecchia P, Staessen JA, Angeli F, de Simone G, Achilli A, Ganau A, Mureddu G, Pede S, Maggioni AP, Lucci D, Reboldi G; Cardio-Sis investigators. Usual versus tight control of systolic blood pressure in non-diabetic patients with hypertension (Cardio-Sis): an open-label randomised trial. Lancet. 2009 Aug 15;374(9689):525-33. doi: 10.1016/S0140-6736(09)61340-4. PMID 19683638
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2022 Nov 18;11(11):CD010315. doi: 10.1002/14651858.CD010315.pub5. PMID 36398903
- [Derived] Saiz LC, Gorricho J, Garjon J, Celaya MC, Erviti J, Leache L. Blood pressure targets for the treatment of people with hypertension and cardiovascular disease. Cochrane Database Syst Rev. 2020 Sep 9;9(9):CD010315. doi: 10.1002/14651858.CD010315.pub4. PMID 32905623